CLINICAL TRIAL: NCT03208595
Title: Endometrial Flora Sampling in Women Undergoing IVF/PGD Treatments
Brief Title: Endometrial Flora in Women Undergoing IVF Treatments
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Deputy Director General for R&D, Tel-Aviv Sourasky Medical Center
Other Study IDs: 0201-17
Record Dates: First submitted 2017-06-26; First posted 2017-07-05 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: Endometrial Flora Characterization in Infertile Women

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bacterial DNA only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Endometrial sampling of a Typical Embryo transfer catheter — no intervention no additional change from unit protocol
  Other Names: no intervention

SUMMARY:
Characterization of the female genital tract microbiome in women undergoing IVF treatment

DETAILED DESCRIPTION:
The primary goal With The purpose of our study is to examine the uterine microbiome by Next-generation sequencing of the bacteria specific regions .

Vaginal and uterine swabs will be taken in different women undergoing IVF /PGD. Novel bacteria and results of taxonomy assignments will be examine to find correlation of uterine flora with IVF and obstetrical outcomes.

The metagenomics approach will be used to seek previously unidentified bacterial species in the human upper genital tract.

ELIGIBILITY:
Inclusion Criteria:

* All undergoning IVF treatment
* Embryo transfer of one Blastocyst

Exclusion Criteria:

* More then one Embryo Transfer
* Recent antibacterial treatment

Ages: 20 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — All infertile women
Study Population: patients undergoing transfer of a single euploid blastocyst .The specimen will be obtaine from the embryo transfer catheter.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
To assess endometrial caracteristicas in fertile and infertile women using next generation sequencing of bacterial identification | 2017-2020
  Type of flora identified by next generation sequencing of bacterial identification
To identify specific endometrial flora in association to faliure of IVF treatment | 2017-2020
  Type of flora identified by NGS
to assess the feasibility of endometrial sampling in women undergoing embryo transfer by a standart transfer cateteher | 2017-2020
  Mode of endometrial sampling

IPD SHARING:
Plan to Share IPD: Undecided